CLINICAL TRIAL: NCT03360084
Title: Systemic Air Embolism After CT-guided Lung Biopsy: Incidence and Risk Factors Assessment
Brief Title: Systemic Air Embolism After CT-guided Lung Biopsy
Acronym: SAE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0326
Record Dates: First submitted 2017-11-23; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Patients Who Underwent Percutaneous Lung Biopsy Under CT Guidance; Patients Who Presented Systemic Air Embolism After Percutaneous Lung Biopsy Under CT Guidance Depicted at the Time of the Procedure on a Whole Thoracic CT
Keywords: CT; Interventional radiology; Lung biopsy; Transthoracic biopsy; Systemic air embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous lung biopsy under CT guidance — Percutaneous lung biopsy under CT guidance

SUMMARY:
Systemic air embolism is traditionally considered as an extremely rare complication of percutaneous lung biopsy. Current literature includes mainly case reports or small case series of SAE. Majority of cases resulted in cardiac and/or neurological symptoms, often causing death. In most reported cases, the diagnosis of systemic air embolism referred to clinical manifestations without radiological diagnosis at the time of the procedure. Hence, its incidence might be underestimated in case of asymptomatic patients. Immediate recognition of air embolism during the procedure has been reported as the main factor to minimize severe complications since specific management of patient can be initiated earlier.

The purpose of this study is to retrospectively assess the incidence of systemic air embolism depicted at the time of the procedure on a whole thoracic CT, systematically performed after transthoracic lung biopsy in a large cohort of consecutive patients. Secondary objectives are to determine possible influencing factors and to evaluate clinical outcomes.

DETAILED DESCRIPTION:
In this retrospective cohort study, all consecutive lung biopsies performed between April 2014 to May 2016 at our department of cardiothoracic interventional radiology were included using the local thoracic biopsy database. Biopsies were scheduled after the weekly multidisciplinary lung cancer meeting approval. Pleural, parietal and mediastinal lesions were excluded due to the absence of intra-parenchymal pathway. Radiofrequency ablation and peripheral nodule marking procedure were also excluded.

A complete retrospective imaging review of the procedures was performed on a PACS workstation by an experienced chest radiologist. Clinical data was also collected from the electronic medical record system.

Variables analyzed were age, sex, spirometry data, emphysema on CT, therapeutics previously done, target lesion characteristics (location, depth, and nodule size and feature), patient position, length of intrapulmonary biopsy path, number of pleural needle passes, biopsy length and number of biopsy passes. Procedural air embolism and other associated complications (hemoptysis and pneumothorax) and their management and consequences (length of hospitalization and additional action) were recorded.

Patient's characteristics with and without air embolism were compared using Student or Wilcoxon rank test for continuous variables and Chi-square or Fisher test for categorical ones. To determine the relative importance of air embolism occurrence influencing factors, multivariate logistic regression analysis was performed on variables according to significance level or clinical coherence. A backward selection was used; the α-to-enter and the α-to-exit were set, respectively, at 0.20 and 0.10. Statistical bilateral significance threshold was set at 5%. Statistical analyses were performed using SAS version 9.1 (SAS Institute, Cary, North Carolina).

ELIGIBILITY:
Inclusion Criteria:

- percutaneous CT guided lung biopsies

Exclusion criteria:

* absence of intra-parenchymal pathway (pleural, parietal or mediastinal lesions)
* radiofrequency ablation
* peripheral nodule marking procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive lung biopsies performed between April 2014 to May 2016 at our department of cardiothoracic interventional radiology were included using the local thoracic biopsy database.
Sampling Method: Non-Probability Sample
Enrollment: 559 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of systemic air embolism | 1 day
  Systemic air embolism was depicted on the CT scan performed on the whole chest in the same position as for the biopsy at the end of the procedure.
  Air embolism was defined as an air collection in the left cardiac cavities or vascular systemic structure, visible in at least two consecutive slices, that was not present on the pre-therapeutic CT

SECONDARY OUTCOMES:
Risk factors of systemic air embolism | 1 day
  Variables were recorded using a retrospective imaging review of the biopsy procedures. Clinical data was also collected from the electronic medical record system.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Monnin-Bares, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France